CLINICAL TRIAL: NCT07154667
Title: Enhancing Cartilaginous Ear Reconstruction - An Institutional Outcomes Study
Brief Title: Evaluation of the Auryzon™ EAR 2.0 System in Ear Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Angelo Leto barone, Craniofacial and Pediatric Plastic Surgeon, Nemours Children's Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000371
Record Dates: First submitted 2025-08-15; First posted 2025-09-04 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Microtia, Congenital; Microtia; Microtia-Anotia; Ear Deformities, Acquired; Ear Deformity External; Ear Malformation; Ear Cartilage
Keywords: microtia; ear reconstruction; craniofacial difference; anotia; plastic surgery; ear defect; ear trauma; ear deficit
MeSH Terms: conditions — Congenital Microtia; Microtia-Anotia; Ear Deformities, Acquired

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AuryzoN™ EAR 2.0 arm (Experimental): Participants in the AuryzoN™ EAR 2.0 arm will receive ear reconstruction surgery using the AuryzoN™ EAR 2.0 device
  Interventions: Procedure: Use of AuryzoN™ EAR 2.0 device
- Hand Carved (Active Comparator): Participants in this arm will receive ear reconstruction surgery using the hand carved technique
  Interventions: Procedure: Hand carving

INTERVENTIONS:
Procedure: Use of AuryzoN™ EAR 2.0 device — AuryzoN™ EAR 2.0 is an investigational non-significant risk device developed to improve cartilage construct shape and stability prior to use in ear reconstructive surgery.
  Arms: AuryzoN™ EAR 2.0 arm
Procedure: Hand carving — Standard hand carving using standard surgical blades will be performed in this intervention arm of the study.
  Arms: Hand Carved

SUMMARY:
This study aims to improve surgical outcomes for children and young adults with ear differences severe secondary to congenital conditions (like microtia, a condition where the ear is underdeveloped), trauma (such as dog bites), or surgical resections secondary to skin cancer. The investigators have developed a novel medical device to shape cartilage into pre-determined shapes that, once assembled, assists the surgeon in creating an anatomically accurate cartilaginous ear framework, reduce surgery time, and minimize wire need. Other factors that might affect the quality of surgical outcomes will be examined in clinical trial participants.

DETAILED DESCRIPTION:
Cartilage-based ear reconstruction addresses congenital anomalies, such as microtia, as well as deformities due to trauma or oncologic resection by replacing like with like tissue. Current technique involves the use of the autologous cartilage as the gold standard and involves harvesting patient's own rib cartilage and carving them into different ear subunits, which are then assembled with numerous steel wires. Challenges of this technique include high operator-dependency due to extensive carving, inconsistent outcomes, prolonged anesthesia, and need for wire or suture fixation, leading to wire extrusion, cartilage resorption, and overall high cost. The previously published prototype device utilized specialized blades to standardize this process. Given the complexity of auricular reconstruction and the suboptimal outcomes by most plastic surgeons globally, there is a pressing need for a standardized, enhanced and accessible method for an accurate ear framework.

If successful, this project has the potential to improve plastic surgeons' technical proficiency in producing anatomically accurate auricular frameworks. Achieving these aims could substantially advance reconstructive clinical techniques in clinical practice and broaden access to satisfactory ear reconstruction beyond the limited number of highly specialized centers. Furthermore, the novel blade design has the potential to reduce the need for wire suturing, while also reducing overall framework production time, anesthesia duration, and costs.

Comparing hand-carved and blade-cut techniques for cadaveric cartilage, the study will enhance understanding of potential differences in resorption rate between these methods. This study aims to: 1. Promote framework production through precise bladecutting, facilitating the construction of cartilaginous ear frameworks while improving outcomes and reducing operative time and costs; 2. Standardize framework production independently of operator skill. 3. Reduce the number of wires required for construct fixation, further contributing to decreased operative time and cost; 4. Minimize the risk of wire extrusion by limiting wires usage during framework production through the novel blade design. 5. Compare differences in framework appearance, stability, time to production, operative time, intraoperative morbidity, and construct resorption within the first year postoperatively when using cadaveric cartilage.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 5-20 years seeking to undergo surgical ear reconstruction or microtia repair under general anesthesia through NCH-FL
* Pre-existing physical deformity of the ear necessitating surgical reconstruction
* Patient of sufficient health to undergo surgery under general anesthesia
* Parental or legally acceptable representative (LAR) permission obtained for inclusion in the study; patient assent obtained where age-appropriate
* Sufficient fluency in English or Spanish to complete patient/parent surveys

Exclusion Criteria:

* Patients who will be ≤4 years old, or ≥21 years old at time of surgery
* Patients with ear deformities do not require surgical correction
* Patient's whose ear reconstruction surgery will be performed somewhere other than Nemours Children's Hospital - Florida
* Patients determined to be in poor health to undergo surgery under general anesthesia
* Parental or LAR permission cannot be obtained, and/or patient of sufficient age and cognitive capacity declines to assent
* Lack of fluency in English or Spanish to complete patient/parent surveys

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the results of patient and parent satisfaction with the constructed ear's shape and appearance and compare the results between the hand-carved cohort and the AuryzoN™ EAR 2.0 cohort using a four-question survey. | From the beginning of the study to the end at 5 years
  Parents and patients (over age 12) will complete a four-question survey asking how much they like: the shape of the new ear, how the new ear looks, how natural the new ear looks, and the new ear overall. Participants will respond to each question with a rating from 1-5, with 1 being "do not like it at all" and 5 being "like it very much". Investigators will compare the responses from the hand-carved cohort and the AuryzoN™ EAR 2.0 cohort to determine which has more favorable outcomes.
Evaluating reduction in operative time between the two techniques. | From the beginning of the study to the end at 5 years
  Compare changes in operative time between participants enrolled in the AuryzoN™ EAR 2.0 arm and the traditional hand-carving arm.
Evaluating reduction in assembly time between the two techniques. | From the beginning of the study to the end at 5 years
  Compare the assembly time of cartilage into the ear construct between the AuryzoN™ EAR 2.0 arm and the hand-carving technique.
Evaluating reduction in wire usage between the two techniques | From the beginning of the study to the end at 5 years
  Compare the amount of wire required for assembly of the ear construct between the Auryzon™ EAR 2.0 arm and the hand-carving technique.
Evaluation of cartilage stability | From the beginning of the study to the end at 5 years
  Assess cartilage framework stability over 12 months post-surgically using photography, measurements, 3D imaging, and histopathological analysis.
Evaluation of resorption rates | From the beginning of the study to the end at 5 years
  Assess resorption rates over 12 months post-surgically using photography, measurements, 3D imaging and histopathological analysis.

SECONDARY OUTCOMES:
Conduct histopathological analysis assessing outcomes of banked allogeneic cartilage between stage 1 and stage 2 surgeries | From the beginning of the study to the end at 5 years
  Cartilage will be banked in participants' groin or supraclavicular region during the six months between stage 1 and stage 2 ear reconstruction surgeries. Investigators will conduct histopathological analysis to assess the quality of the banked cartilage when it is recovered for use in the stage 2 surgery. This pathological analysis of the banked cartilage will be performed by using Hematoxylin & Eosin (H&E) staining and evaluating chondrocytes and extracellular matrix for signs of inflammatory response or rejection.
Assessing any changes to the dimensions of the banked cartilage when it is retrieved for stage 2 reconstruction surgery. | From the beginning of the study to the end at 5 years
  Surgeons will measure the dimensions of the cartilage before banking at the end of the stage 1 surgery and after retrieving the banked cartilage during the stage 2 surgery. Investigators will compare the dimensions of the cartilage before and after banking to determine whether there are any signing or warping or resorption

CONTACTS AND LOCATIONS:
Overall Officials: Angelo A Leto Barone, MD, Principal Investigator — Nemours Children's Hospital, Florida
Locations (1):
- Nemours Children's Hospital, Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagata S. A new method of total reconstruction of the auricle for microtia. Plast Reconstr Surg. 1993 Aug;92(2):187-201. doi: 10.1097/00006534-199308000-00001. PMID 8337267
- [Background] Tanzer RC. Microtia--a long-term follow-up of 44 reconstructed auricles. Plast Reconstr Surg. 1978 Feb;61(2):161-6. doi: 10.1097/00006534-197802000-00001. PMID 622405
- [Background] Su-Genyk P, Quatela O, Quatela V. Our Evolution of Approaches to Microtia Reconstruction. Facial Plast Surg Clin North Am. 2024 Feb;32(1):105-125. doi: 10.1016/j.fsc.2023.09.002. PMID 37981407
- See also: Nemours Plastic Surgery Website — https://www.nemours.org/services/pediatric-plastic-surgery.html